CLINICAL TRIAL: NCT07004556
Title: The Effect of Laparoscopic Sleeve Gastrectomy on Blood Phoenixin-14 Levels: A Prospective Cohort Study
Brief Title: The Effect of Laparoscopic Sleeve Gastrectomy on Blood Phoenixin-14 Levels
Acronym: Morbid Obesity
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Mehmet Buğra Bozan, Professor, Associate (MD), Elazıg Fethi Sekin Sehir Hastanesi
Other Study IDs: 2025/9-9; 2025/9-9 (Registry Identifier: ELAZIĞ FETHİ SEKİN ŞEHİR HASTANESİ Girişimsel Olmayan Araştırmalar Etik Kurulu)
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Obesity, Morbid; Obesity and Overweight
Keywords: Severe Obesity; Laparoscopic Sleeve Gastrectomy; Phoenixin-14; Obesity Surgery
MeSH Terms: conditions — Obesity, Morbid; Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Selective Laparoscopic Sleeve Gastrectomy Patients: Preoperative and postoperative blood samples obtained from the patients
  Interventions: Diagnostic Test: Preoperative blood sampling for determining Phoenixin 14 levels; Diagnostic Test: Postoperative blood sampling for determining Phoenixin 14 levels

INTERVENTIONS:
Diagnostic Test: Preoperative blood sampling for determining Phoenixin 14 levels — In addition to routine blood draws for pre-operative preparations, 5 ml of blood will be collected.
Diagnostic Test: Postoperative blood sampling for determining Phoenixin 14 levels — In addition to routine blood draws for postoperative controls, 5 ml of blood will be collected.

SUMMARY:
Obesity is a major global health concern with a rising prevalence and numerous associated comorbidities. For the treatment of severe obesity, bariatric surgery stands as the most effective procedure. Bariatric and metabolic surgical procedures are applied even in the absence of comorbidities, particularly in patients with Type-III obesity and above. Currently, the most commonly performed bariatric metabolic surgical procedures are Laparoscopic Sleeve Gastrectomy (LSG) and Roux-en-Y gastric bypass.

Animal studies have shown that phoenixin (PNX) in the paraventricular, arcuate, and solitary tract nuclei contributes to regulating food intake, and its intracerebral administration in rats increased food intake.

The aim of this study is to investigate whether PNX-14 levels change before and after LSG in patients undergoing the procedure for severe obesity, given the potential association of PNX-14 with obesity and insulin resistance through its influence on the appetite center in metabolism.

DETAILED DESCRIPTION:
Introduction Obesity is a major global health concern with a rising prevalence and numerous associated comorbidities. In 2022, approximately 2.5 billion adults (aged 18 and over) were overweight (BMI between 25 kg/m² and 30 kg/m²), with 890 million of them categorized as obese (BMI ≥ 30 kg/m²).

For the treatment of severe obesity, bariatric surgery stands as the most effective procedure. Bariatric and metabolic surgical procedures are applied even in the absence of comorbidities, particularly in patients with Type-III obesity and above. Various bariatric metabolic surgical techniques have been developed for this purpose. Currently, the most commonly performed bariatric metabolic surgical procedures are Laparoscopic Sleeve Gastrectomy (LSG) and Roux-en-Y gastric bypass.

Animal studies have shown that phoenixin (PNX) in the paraventricular, arcuate, and solitary tract nuclei contributes to regulating food intake, and its intracerebral administration in rats increased food intake. A study by Cundubey et al. in women with polycystic ovary syndrome (PCOS) demonstrated significantly increased serum PNX-14 levels in obese PCOS patients. PNX is not only expressed and secreted by the central nervous system but also by peripheral tissues such as the heart, adipose tissue, pancreas, and stomach. This suggests that PNX-14 plays a crucial role in appetite regulation and energy intake control via the central nervous system.

The aim of this study is to investigate whether PNX-14 levels change before and after LSG in patients undergoing the procedure for severe obesity, given the potential association of PNX-14 with obesity and insulin resistance through its influence on the appetite center in metabolism.

Material-Methods This study is designed as a cross-sectional prospective study. The goal is to include patients who present to the General Surgery Clinic at Elazığ Fethi Sekin City Hospital for severe obesity and are scheduled for Laparoscopic Sleeve Gastrectomy (LSG) as their primary surgery.

In addition to routine pre-operative blood tests, 5 ml of blood will be collected from patients. Another 5 ml will be collected in yellow-capped biochemistry tubes along with routine complete blood count measurements taken for post-operative control. The study will analyze plasma phoenixin-14 (PNX-14) levels both before and after the surgery.

Using the G*power 3.10 program for repeated measures t-tests, a sample size of at least 36 patients was determined to be appropriate to achieve 90% power with an alpha error probability of 0.05 and a medium Cohen's effect size.

Hypotheses H0 (Null Hypothesis): There is no relationship between LSG performed for severe obesity and the change in pre-operative and post-operative plasma phoenixin-14 (PNX-14) levels.

H1 (Alternative Hypothesis): There is a relationship between LSG performed for severe obesity and the change in pre-operative and post-operative blood PNX-14 levels.

Research Budget The research budget will be covered by the principal investigator. Inclusion Criteria Patients aged 18-65 years. Patients with severe obesity (Body Mass Index (BMI) ≥ 40 kg/m²) with no additional comorbidities (Type III, Type IV, and Type V obesity) who are scheduled for primary LSG.

Patients who consent to participate in the study. Exclusion Criteria Patients who do not consent to participate in the study. Patients scheduled for primary obesity surgery other than LSG (e.g., Single Anastomosis Gastric Bypass, Roux-en-Y Gastric Bypass, Transit Bipartition, Single Anastomosis Sleeve Ileal Bypass, Single Anastomosis Duodeno-intestinal Bypass, Duodenal Switch).

Patients with a BMI ≥ 35 kg/m² with associated medical problems (e.g., Diabetes Mellitus, Asthma, Chronic Obstructive Pulmonary Disease, Ischemic Heart Disease, Hypertension).

Patients with a BMI ≤ 35 kg/m² who do not have a surgical indication. Data Collection Tools/Methods

Patient demographics and anthropometrics: Age, gender, height, body weight, and BMI will be recorded. The severity of obesity will be classified based on BMI values:

BMI = Body Weight (kilograms) / (Height x Height) (meters x meters)

Obesity Severity based on BMI (1,2):

BMI ≥ 18 - < 25 kg/m² → Normal BMI ≥ 25 - < 30 kg/m² → Overweight BMI ≥ 30 - < 35 kg/m² → Class I Obesity BMI ≥ 35 - < 40 kg/m² → Class II Obesity BMI ≥ 40 - < 50 kg/m² → Class III Obesity BMI ≥ 50 - < 60 kg/m² → Class IV Obesity BMI ≥ 60 kg/m² → Class V Obesity Blood PNX-14 Levels: In addition to routine blood draws for pre-operative preparations, 5 ml of blood will be collected. Another 5 ml will be collected in a yellow biochemistry tube on the 1st post-operative day, in addition to the routine complete blood count for control purposes.

Samples will be centrifuged at 4000 rpm for approximately 10 minutes at the Elazığ Fethi Sekin City Hospital Biochemistry Laboratory and stored at -20 degrees Celsius until the analysis day.

Once all samples are collected, they will be thawed at room temperature and analyzed using the microELISA method with a kit provided by the researchers. The analysis will be performed by Assoc. Prof. Dr. Hakan Ayyıldız at the Elazığ Fethi Sekin City Hospital Biochemistry Laboratory, adhering to the reagent manufacturer's methodology.

Reaction washes will be performed with a Combiwash-Human device, and absorbance measurements will be taken using a Chromate 4300 Microplate Reader (Awareness Technology, Palm City, USA) at 450 nm. Results will be recorded in an Excel sheet containing patient demographic data.

Statistical Method(s) to be Used Data analysis will be performed using IBM Statistical Analysis for Social Sciences (SPSS) version 20 statistical package program. The Shapiro-Wilk test will be used to assess the normality of numerical data distribution. Numerical data will be expressed as mean ± standard deviation (SD) (minimum - maximum values) or median (95% Confidence Interval), depending on their conformity to normal distribution. Categorical data will be presented as numbers (n) and percentages (%).

For comparing plasma PNX-14 levels, either the paired sample t-test or the Wilcoxon Rank test will be used. A pre-operative and post-operative ROC analysis will be conducted to determine a cut-off value for PNX-14 levels. A probability value of p < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years.
* Patients with severe obesity (Body Mass Index (BMI) ≥ 40 kg/m²) with no additional comorbidities (Type III, Type IV, and Type V obesity) who are scheduled for primary LSG.
* Patients who consent to participate in the study.

Exclusion Criteria:

* Patients who do not consent to participate in the study.
* Patients scheduled for primary obesity surgery other than LSG (e.g., Single Anastomosis Gastric Bypass, Roux-en-Y Gastric Bypass, Transit Bipartition, Single Anastomosis Sleeve Ileal Bypass, Single Anastomosis Duodeno-intestinal Bypass, Duodenal Switch).
* Patients with a BMI ≥ 35 kg/m² with associated medical problems (e.g., Diabetes Mellitus, Asthma, Chronic Obstructive Pulmonary Disease, Ischemic Heart Disease, Hypertension).
* Patients with a BMI ≤ 35 kg/m² who do not have a surgical indication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe obesity patients scheduled for selective laparoscopic sleeve gastrectomy who have no associated medical problems
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Laparoscopic Sleeve Gastrectomy effects blood Phoenixin 14 levels | June 01,2025-October 01,2025
  Phoenixin 14 blood levels can be effected by surgical intervention for severe obesity (laparoscopic sleeve gastrectomy)

CONTACTS AND LOCATIONS:
Locations (1):
- Elazığ Fethi Sekin City Hospital, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Prinz P, Scharner S, Friedrich T, Schalla M, Goebel-Stengel M, Rose M, Stengel A. Central and peripheral expression sites of phoenixin-14 immunoreactivity in rats. Biochem Biophys Res Commun. 2017 Nov 4;493(1):195-201. doi: 10.1016/j.bbrc.2017.09.048. Epub 2017 Sep 11. PMID 28911868
- [Background] Akdu S, Can U, Polat E. Investigation of serum phoenixin levels in patients with hypertension. Rev Assoc Med Bras (1992). 2022 Jun 24;68(6):814-819. doi: 10.1590/1806-9282.20220153. eCollection 2022. PMID 35766697
- [Background] Cundubey CR, Cam SD. Serum Phoenixin-14 levels of women with polycystic ovary syndrome increase proportionally with BMI. Eur Rev Med Pharmacol Sci. 2023 Apr;27(8):3519-3525. doi: 10.26355/eurrev_202304_32125. PMID 37140302
- [Background] Mukherjee K, Unniappan S. Mouse gastric mucosal endocrine cells are sources and sites of action of Phoenixin-20. Peptides. 2021 Jul;141:170551. doi: 10.1016/j.peptides.2021.170551. Epub 2021 Apr 17. PMID 33862165
- [Background] Schalla M, Prinz P, Friedrich T, Scharner S, Kobelt P, Goebel-Stengel M, Rose M, Stengel A. Phoenixin-14 injected intracerebroventricularly but not intraperitoneally stimulates food intake in rats. Peptides. 2017 Oct;96:53-60. doi: 10.1016/j.peptides.2017.08.004. Epub 2017 Aug 24. PMID 28844870
- [Background] Han Y, Jia Y, Wang H, Cao L, Zhao Y. Comparative analysis of weight loss and resolution of comorbidities between laparoscopic sleeve gastrectomy and Roux-en-Y gastric bypass: A systematic review and meta-analysis based on 18 studies. Int J Surg. 2020 Apr;76:101-110. doi: 10.1016/j.ijsu.2020.02.035. Epub 2020 Mar 6. PMID 32151750
- [Background] https://bmjpublichealth.bmj.com/lookup/doi/10.1136/bmjph-2023-000245
- [Background] Kirkil C, Aygen E, Korkmaz MF, Bozan MB. QUALITY OF LIFE AFTER LAPAROSCOPIC SLEEVE GASTRECTOMY USING BAROS SYSTEM. Arq Bras Cir Dig. 2018 Aug 16;31(3):e1385. doi: 10.1590/0102-672020180001e1385. PMID 30133677
- [Background] https://www.who.int/news-room/fact-sheets/detail/obesity-and-overweight
- [Background] Kassir R, Debs T, Blanc P, Gugenheim J, Ben Amor I, Boutet C, Tiffet O. Complications of bariatric surgery: Presentation and emergency management. Int J Surg. 2016 Mar;27:77-81. doi: 10.1016/j.ijsu.2016.01.067. Epub 2016 Jan 22. PMID 26808323
- [Background] Eisenberg D, Shikora SA, Aarts E, Aminian A, Angrisani L, Cohen RV, de Luca M, Faria SL, Goodpaster KPS, Haddad A, Himpens JM, Kow L, Kurian M, Loi K, Mahawar K, Nimeri A, O'Kane M, Papasavas PK, Ponce J, Pratt JSA, Rogers AM, Steele KE, Suter M, Kothari SN. 2022 American Society of Metabolic and Bariatric Surgery (ASMBS) and International Federation for the Surgery of Obesity and Metabolic Disorders (IFSO) Indications for Metabolic and Bariatric Surgery. Obes Surg. 2023 Jan;33(1):3-14. doi: 10.1007/s11695-022-06332-1. PMID 36336720
- [Background] Purnell JQ. Definitions, Classification, and Epidemiology of Obesity. 2023 May 4. In: Feingold KR, Adler RA, Ahmed SF, Anawalt B, Blackman MR, Chrousos G, Corpas E, de Herder WW, Dhatariya K, Dungan K, Hamilton E, Hofland J, Jan de Beur S, Kalra S, Kaltsas G, Kapoor N, Kim M, Koch C, Kopp P, Korbonits M, Kovacs CS, Kuohung W, Laferrere B, Levy M, McGee EA, McLachlan R, Muzumdar R, Purnell J, Rey R, Sahay R, Shah AS, Sperling MA, Stratakis CA, Trence DL, Wilson DP, editors. Endotext [Internet]. South Dartmouth (MA): MDText.com, Inc.; 2000-. Available from http://www.ncbi.nlm.nih.gov/books/NBK279167/ PMID 25905390